CLINICAL TRIAL: NCT02062710
Title: Antitussive Effect of a Naturally Flavored, Multi-Component Syrup Containing Diphenhydramine, Compared With Dextromethorphan and Placebo
Brief Title: Antitussive Effect of a Naturally Flavored Syrup Containing Diphenhydramine, Compared With Dextromethorphan and Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Peter Dicpinigaitis, Principal Investigator, Montefiore Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MMC-IRB-13-10-170
Record Dates: First submitted 2014-01-31; First posted 2014-02-14 (Estimated); Results first posted 2015-04-28 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Cough Reflex Sensitivity
Keywords: cough; cough reflex; capsaicin; diphenhydramine; phenylephrine; dextromethorphan; placebo
MeSH Terms: conditions — Cough | interventions — Diphenhydramine; Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A, B, then C (Experimental): Subjects received the following: Period 1: single oral dose of diphenhydramine 25 mg and phenylephrine 10 mg, in naturally-flavored cocoa syrup (treatment A). Period 2: dextromethorphan syrup 30 mg (treatment B); Period 3: placebo liquid, dextrose in water, 20 mL (treatment C).
  Intervention: capsaicin cough challenge testing 2 hours after study drug ingestion.Each dosing period separated by 1-2 day washout period.
  Interventions: Drug: diphenhydramine/phenylephrine/cocoa; dextromethorophan; placebo; Drug: diphenhydramine/phenylephrine/cocoa; placebo; dextromethorphan; Drug: dextromethorphan; diphenhydramine/phenylephrine/cocoa; placebo; Drug: dextromethorophan; placebo; diphenhydramine/phenylephrine/cocoa; Drug: placebo; diphenhydramine/phenylephrine/cocoa; dextromethorphan; Drug: placebo; dextromethorphan; diphenhydramine/phenylephrine/cocoa
- A, C, then B (Experimental): Subjects received the following: Period 1: single oral doce of diphenhydramine 25 mg and phenylephrine 10 mg, in naturally-flavored cocoa syrup (treatment A); Period 2: placebo liquid, dextrose in watwer, 20 mL (treatment C); Period 3: dextromethorphan syrup 30 mg (treatment B).
  Intervention: capsaicin cough challenge testing 2 hours after study drug ingestion.Each dosing period separated by 1-2 day washout period.
  Interventions: Drug: diphenhydramine/phenylephrine/cocoa; dextromethorophan; placebo; Drug: diphenhydramine/phenylephrine/cocoa; placebo; dextromethorphan; Drug: dextromethorphan; diphenhydramine/phenylephrine/cocoa; placebo; Drug: dextromethorophan; placebo; diphenhydramine/phenylephrine/cocoa; Drug: placebo; diphenhydramine/phenylephrine/cocoa; dextromethorphan; Drug: placebo; dextromethorphan; diphenhydramine/phenylephrine/cocoa
- B, A, then C (Experimental): Subjects received the following: Period 1: dextromethorphan syrup 30 mg (treatment B); Period 2: single dose of oral diphenhydramine 25 mg and phenylephrine 10 mg, in a naturally-flavored cocoa syrup (treatment A); Period 3: placebo liquid, dextrose in water, 20 mL (treatment C). Intervention: capsaicin cough challenge testing 2 hours after study drug ingestion. Each dosing period separated by 1-2 day washout period.
  Interventions: Drug: diphenhydramine/phenylephrine/cocoa; dextromethorophan; placebo; Drug: diphenhydramine/phenylephrine/cocoa; placebo; dextromethorphan; Drug: dextromethorphan; diphenhydramine/phenylephrine/cocoa; placebo; Drug: dextromethorophan; placebo; diphenhydramine/phenylephrine/cocoa; Drug: placebo; diphenhydramine/phenylephrine/cocoa; dextromethorphan; Drug: placebo; dextromethorphan; diphenhydramine/phenylephrine/cocoa
- B, C, then A (Experimental): Subjects received the following: Period 1: dextromethorphan 30 mg syrup (treatment B); Period 2: placebo liquid, dextrose in water, 20 mL (treatment C); Period 3: single dose of oral diphenhydramine 25 mg and phenylephrine 10 mg in a naturally-flavored cocoa syrup (treatment A).
  Intervention: capsaicin cough challenge testing 2 hours after study drug ingestion. Each dosing period separated by 1-2 day washout period.
  Interventions: Drug: diphenhydramine/phenylephrine/cocoa; dextromethorophan; placebo; Drug: diphenhydramine/phenylephrine/cocoa; placebo; dextromethorphan; Drug: dextromethorphan; diphenhydramine/phenylephrine/cocoa; placebo; Drug: dextromethorophan; placebo; diphenhydramine/phenylephrine/cocoa; Drug: placebo; diphenhydramine/phenylephrine/cocoa; dextromethorphan; Drug: placebo; dextromethorphan; diphenhydramine/phenylephrine/cocoa
- C, A, then B (Experimental): Subjects received the following: Period 1: placebo liquid, dextrose in water, 20 mL (treatment C); Period 2: a single oral dose of diphenhydramine 25 mg and phenylephrine 10 mg in a naturally-flavored cocoa syrup (treatment A); Period 3: dextromethorphan 30 mg syrup (treatment B). Intervention: capsaicin cough challenge testing 2 hours after study drug ingestion. Each dosing period separated by 1-2 day washout period.
  Interventions: Drug: diphenhydramine/phenylephrine/cocoa; dextromethorophan; placebo; Drug: diphenhydramine/phenylephrine/cocoa; placebo; dextromethorphan; Drug: dextromethorphan; diphenhydramine/phenylephrine/cocoa; placebo; Drug: dextromethorophan; placebo; diphenhydramine/phenylephrine/cocoa; Drug: placebo; diphenhydramine/phenylephrine/cocoa; dextromethorphan; Drug: placebo; dextromethorphan; diphenhydramine/phenylephrine/cocoa
- C, B, then A (Experimental): Subjects received the following: Period 1: placebo liquid, dextrose in water, 20 mL (treatment C); Period 2: dextromethorphan 30 mg syrup (treatment B); Period 3: a single oral dose of diphenhydramine 25 mg and phenylephrine 10 mg in a naturally-flavored cocoa syrup (treatment A). Intervention: capsaicin cough challenge testing 2 hours after study drug ingestion. Each dosing period separated by 1-2 day washout period.
  Interventions: Drug: diphenhydramine/phenylephrine/cocoa; dextromethorophan; placebo; Drug: diphenhydramine/phenylephrine/cocoa; placebo; dextromethorphan; Drug: dextromethorphan; diphenhydramine/phenylephrine/cocoa; placebo; Drug: dextromethorophan; placebo; diphenhydramine/phenylephrine/cocoa; Drug: placebo; diphenhydramine/phenylephrine/cocoa; dextromethorphan; Drug: placebo; dextromethorphan; diphenhydramine/phenylephrine/cocoa

INTERVENTIONS:
Drug: diphenhydramine/phenylephrine/cocoa; dextromethorophan; placebo — diphenhydramine 25 mg and phenylephrine 10 mg; dextromethorphan 30 mg; placebo.
Drug: diphenhydramine/phenylephrine/cocoa; placebo; dextromethorphan — diphenhydramine 25 mg and phenylephrine 10 mg; placebo; dextromethorphan 30 mg.
Drug: dextromethorphan; diphenhydramine/phenylephrine/cocoa; placebo — dextromethorphan 30 mg; diphenhydramine 25 mg and phenylephrine 10 mg; placebo
Drug: dextromethorophan; placebo; diphenhydramine/phenylephrine/cocoa — dextromethorphan 30 mg; placebo; diphenhydramine 25 mg and phenylephrine 10 mg
Drug: placebo; diphenhydramine/phenylephrine/cocoa; dextromethorphan — placebo; diphenhydramine 25 mg and phenylephrine 10 mg; dextromethorphan 30 mg
Drug: placebo; dextromethorphan; diphenhydramine/phenylephrine/cocoa — placebo; dextromethorphan 30 mg; diphenhydramine 25 mg and phenylephrine 10 mg

SUMMARY:
The purpose of this study is to evaluate the antitussive (cough-suppressing) effects of two liquid medications: a combination of diphenhydramine and phenylephrine in a naturally cocoa flavoring, and, dextromethorphan syrup, compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult nonsmokers
* onset of acute, viral upper respiratory tract infection (common cold) within 72 hours of enrollment

Exclusion Criteria:

* smokers
* history of asthma or other respiratory disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Einstein Division/Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Dicpinigaitis PV, Dhar S, Johnson A, Gayle Y, Brew J, Caparros-Wanderley W. Inhibition of cough reflex sensitivity by diphenhydramine during acute viral respiratory tract infection. Int J Clin Pharm. 2015 Jun;37(3):471-4. doi: 10.1007/s11096-015-0081-8. Epub 2015 Feb 12. PMID 25673148

RESULTS

PARTICIPANT FLOW:
Groups:
- Diphenhydramine/Phen/Cocoa, Dextromethorphan, Then Placebo: Diphenhydramine 25 mg, phenylephrine 10 mg, in naturally-flavored cocoa syrup; then dextromethorphan 30 mg; then placebo.
  Intervention: capsaicin cough challenge testing 2 hours after study drug ingestion.
  Washout 1-2 days between each of the 3 dosing periods.
- Diphenhydramine/Phenylephrine/Cocoa, Then Placebo, Then Dextro: diphenhydramine 25 mg and phenylephrine 10 mg; then placebo; then dextromethorphan 30 mg.
  Intervention: capsaicin cough challenge testing after study drug ingestion
- Dextromethorphan, Diphenhydramine/Phenylephrine/Cocoa, Then pl: dextromethorphan 30 mg, then diphenhydramine/phenylephrine/cocoa, then placebo. Intervention: capsaicin cough challeneg 2 hours after study drug ingestion
- Dextromethorphan, Placebo, Then Diphenhydramine/Phenylephrine/: dextromethorphan 30 mg, then placebo, then diphenhydramine 25 mg and phenylephrine 10 mg.
  Intervention: capsaicin cough challenge 2 hours after study drug ingestion. Washout period 1-2 days between each of the 3 dosing periods
- Placebo, Diphenhydramine/Phenylephrine/Cocoa, Then Dextrometho: placebo, then diphenhydramine 25 mg and phenylephrine 10 mg, then dextromethorphan 30 mg.
  Intervention: capsaicin cough challenge 2 hours after study drug administration.
  Washout period 1-2 days after each of the 3 dosing periods
- Placebo, Dextromethorphan, Then Diphenhydramine/Phenylephrine/: placebo, then dextromethorphan 30 mg, then diphenhydramine 25 mg and phenylephrine 10 mg.
  Intervention: capsaicin cough challenge 2 hours after study drug administration.
  Washout period 1-2 days after each of the 3 dosing periods.
Period: Overall Study
Arm/Group | Diphenhydramine/Phen/Cocoa, Dextromethorphan, Then Placebo | Diphenhydramine/Phenylephrine/Cocoa, Then Placebo, Then Dextro | Dextromethorphan, Diphenhydramine/Phenylephrine/Cocoa, Then pl | Dextromethorphan, Placebo, Then Diphenhydramine/Phenylephrine/ | Placebo, Diphenhydramine/Phenylephrine/Cocoa, Then Dextrometho | Placebo, Dextromethorphan, Then Diphenhydramine/Phenylephrine/
Started | 3 (3 of total 22 subjects randomized to receive the 3 study drugs in this particular sequence) | 4 (4 of the total 22 subjects randomized to receive the 3 study drugs in this particular sequence) | 5 (5 of total of 22 subjects randomized to receive the 3 study drugs in this particular sequence) | 3 (3 of 22 subjects randomized to receive the 3 study drugs in this particular sequence) | 3 (3 of 22 subjects randomized to receive the 3 study drugs in this aprticular sequence) | 4 (4 of 22 subjects randomized to receive the 3 study drugs in this particular sequence)
Completed | 3 | 4 | 5 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Diphenhydramine/Phenylephrine/Cocoa, Dextromethorphan,Placebo: Diphenhydramine 25 mg, phenylephrine 10 mg, in naturally-flavored cocoa syrup; dextromethorphan; placebo.
  Intervention: capsaicin cough challenge testing 2 hours after study drug ingestion.
  Phenylephrine: 10 mg dose phenylephrine
  Diphenhydramine: 25 mg dose diphenhydramine
  Dextromethorphan: 30 mg dose dextromethorphan
Arm/Group | Diphenhydramine/Phenylephrine/Cocoa, Dextromethorphan,Placebo
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Cough Reflex Sensitivity to Capsaicin
Description: increase in C5 (decrease in cough reflex sensitivity). Capsaicin cough challenge involves subjects breathing in incremental doubling concentrations of aerosolized capsaicin, 1 minute apart, until the concentration of capsaicin (micromolar) inducing 5 or more coughs (C5) is reached.
Time Frame: 2 hours after study drug administration
Measure: Mean (Standard Error); unit: log C5 (uM)
Groups:
- Diphenhydramine/Phenylephrine/Cocoa: Diphenhydramine 25 mg, phenylephrine 10 mg, in naturally-flavored cocoa syrup. Intervention: capsaicin cough challenge testing 2 hours after study drug ingestion.
  Phenylephrine: 10 mg dose phenylephrine
  Diphenhydramine: 25 mg dose diphenhydramine
- Dextromethorphan: Dextromethorphan syrup, 30 mg dose. Intervention: capsaicin cough challenge testing 2 hours after study drug ingestion.
  Dextromethorphan: 30 mg dose dextromethorphan
- Placebo: placebo liquid, dextrose in water, 20 mL
Arm/Group | Diphenhydramine/Phenylephrine/Cocoa | Dextromethorphan | Placebo
Number analyzed (Participants) | 22 | 22 | 22
log C5 (uM) | 0.97 (0.16) | 0.80 (0.18) | 0.57 (0.16)

ADVERSE EVENTS:
Arm/Group | Diphenhydramine/Phenylephrine/Cocoa | Dextromethorphan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No